CLINICAL TRIAL: NCT05479617
Title: Personalised Prediction of Disease Course in Ulcerative Colitis Using Multimodal Machine Learning - Part of the Presager Project
Acronym: Presager II
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Bobby Lo, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-21020965
Record Dates: First submitted 2022-06-29; First posted 2022-07-29 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Deep learning model — Use of deep learning model to predict individual patients disease course

SUMMARY:
In patients achieving clinical remission following a flare, artificial intelligence can reliably predict a new flare within the next 12 months utilizing clinical and objective information at day 0 and week 8.

Secondary endpoints:

* An artificial intelligence model's precision in predicting a new flare within 2 and 3 years
* An artificial intelligence model's precision to rule out patients who will not experience a new flare within 1, 2 and 3 year

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* Diagnosis of UC for at least 1 year
* Relapse due to UC.
* First endoscopic and histological evaluation of the flare Exclusion criteria
* Well-founded doubt that the flare is due to other than the patients UC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort of a total of 400 UC patients with an active flare
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Flare I | within 1 year
  Evaluate the accuracy in predicting a flare within 1 year after the patient's initial flare using machine learning methods.

SECONDARY OUTCOMES:
Flare II | within 2 years
  Evaluate the accuracy in predicting a flare within 2 years, after the patient's initial flare, using machine learning methods.
Flare III | within 3 years
  Evaluate the accuracy in predicting a flare within 3 years, after the patient's initial flare, using machine learning methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrounit, medical section, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The description is in Danish — https://www.hvidovrehospital.dk/cph-ibd/forskning/projekter/Sider/PRESAGER.aspx